CLINICAL TRIAL: NCT07314749
Title: Physician-Nurse Intervention With An Intelligent System for Hypoglycemia in Type 2 Diabetes Patients
Brief Title: 2025 Hypoglycemia Early-Warning and Physician-Nurse Collaborative Management Trial in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Xiling Hu, Chief Nurse, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR-44-25-024286; 2025A1515012706 (Other Grant/Funding Number: Guangdong Basic and Applied Basic Research Foundation); A2024530 (Other Grant/Funding Number: Medical Scientific Research Foundation of Guangdong Province of China); YHJH202404 (Other Grant/Funding Number: 3rd Affiliated Hospital of Sun Yat-sen University, Clinical Research Program); 72204277 (Other Grant/Funding Number: National natural science foundation of China); YJYZ202304 (Other Grant/Funding Number: Nursing innovation development research project)
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Hypoglycemia; Intensive Insulin Therapy; Physician-nurse collaboration; Risk early-warning system; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Physician-Nurse Collaborative Intervention Guided by Intelligent Hypoglycemia Risk Early-Warning System
- Control Group (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Physician-Nurse Collaborative Intervention Guided by Intelligent Hypoglycemia Risk Early-Warning System — Participants in this arm will receive standard insulin pump therapy combined with a physician-nurse collaborative intervention guided by an Intelligent Hypoglycemia Risk Early-Warning System. The intervention includes individualized insulin dose adjustment, intensified glucose monitoring, risk-stratified hypoglycemia prevention strategies, targeted education, and nurse follow-up based on real-time risk alerts.
  Arms: Intervention Group
Other: Usual Care — Participants in this arm will receive standard insulin pump therapy and usual nursing care according to routine hospital practice, without the use of the Intelligent Hypoglycemia Risk Early-Warning System or the physician-nurse collaborative intervention.
  Arms: Control Group

SUMMARY:
The goal of this clinical study is to learn whether a physician-nurse collaborative intervention guided by an Intelligent Hypoglycemia Risk Early-Warning System can reduce hypoglycemia and improve glycemic control in hospitalized adults with type 2 diabetes receiving intensive insulin pump therapy. The study also aims to understand how risk-stratified management influences the time needed to reach glycemic targets.

The main questions this study aims to answer are:

1. Does the physician-nurse collaborative intervention reduce the incidence of hypoglycemia, particularly level 2 and symptomatic hypoglycemia?
2. Does this intervention help patients reach their glycemic targets sooner during intensive insulin pump therapy?
3. What differences in outcomes are observed between patients classified as high-risk and low-risk by the Intelligent Hypoglycemia Risk Early-Warning System?

Participants will:

1. Receive either standard insulin pump therapy alone or insulin pump therapy combined with the physician-nurse collaborative intervention
2. Undergo hypoglycemia risk assessment using the Intelligent Early-Warning System
3. Receive individualized insulin dose adjustments, intensified glucose monitoring, and tailored hypoglycemia education based on their risk category
4. Be monitored for hypoglycemic events and time to achieve glycemic targets during hospitalization This study will compare the collaborative intervention with standard care to evaluate its effectiveness in preventing hypoglycemia and accelerating glycemic stabilization among hospitalized patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus.
* Age 18 years or older.
* Hospitalized for 3 days or longer.
* Receiving continuous subcutaneous insulin infusion (CSII) therapy during hospitalization.

Exclusion Criteria:

* Acute diabetic complications (e.g., diabetic ketoacidosis, hyperosmolar hyperglycemic state).
* Severe cardiovascular or cerebrovascular disease, hepatic dysfunction, or renal dysfunction.
* Malignant tumors.
* Severe cognitive impairment or psychiatric disorders that prevent cooperation.
* Premature discontinuation of CSII therapy due to non-glycemic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1255 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypoglycemia | From the date of randomization until hospital discharge, assessed up to 14 days.
  The proportion of participants experiencing hypoglycemia, defined as blood glucose < 3.9 mmol/L. Hypoglycemia will be further classified into level 1, level 2, level 3, symptomatic, and asymptomatic categories based on international clinical criteria.

SECONDARY OUTCOMES:
Time to Glycemic Target | From the date of randomization until achievement of predefined glycemic targets, assessed up to 14 days.
  Time required for participants to reach predefined glycemic targets during insulin pump therapy. Glycemic targets are defined as fasting blood glucose 4.4-7.0 mmol/L and 2-hour postprandial glucose < 10.0 mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive personal health information and is restricted by institutional and ethical requirements.